CLINICAL TRIAL: NCT02354222
Title: Confirmatory Study of MT-2412 in Japanese Patients With Type 2 Diabetes (Add-on Study of Teneligliptin in Patients With Inadequate Glycemic Control on Canagliflozin)
Brief Title: Confirmatory Study of MT-2412 in Japanese Patients With Type 2 Diabetes (Add-on Study of Teneligliptin)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-2412-J02
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: MT-2412; MP-513; TA-7284; Teneligliptin; Canagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teneligliptin + Canagliflozin (Experimental): Patients receive Teneligliptin for 24 weeks in combination with Canagliflozin.
  Interventions: Drug: Canagliflozin; Drug: Teneligliptin
- Placebo + Canagliflozin (Placebo Comparator): Patients receive placebo for 24 weeks in combination with Canagliflozin.
  Interventions: Drug: Canagliflozin; Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin
  Other Names: Canaglu, TA-7284
Drug: Teneligliptin
  Other Names: Tenelia, MP-513
  Arms: Teneligliptin + Canagliflozin
Drug: Placebo
  Arms: Placebo + Canagliflozin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of co-administration of Canagliflozin (TA-7284) and Teneligliptin (MP-513) once daily for 24 weeks in Japanese patients with Type 2 diabetes mellitus who are receiving treatment with Canagliflozin and have inadequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are 20 - 75 years old
* HbA1c of ≥7.0% and <10.5%
* FPG of ≤ 270 mg/dL
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 8 weeks before run-in period

Exclusion Criteria:

* Patients with type I diabetes, diabetes mellitus resulting from pancreatic disorder, or secondary diabetes
* Patients with serious diabetic complications
* Patients with hereditary glucose-galactose malabsorption or primary renal glucosuria
* Patients with Class III/IV heart failure symptoms according to New York Heart Association (NYHA) functional classification
* Patients with severe hepatic disorder or severe renal disorder.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, M.D., Study Director — Tokyo University; Kazuoki Kondo, M.D., Study Director — Tanabe Pharma Corporation
Locations (3):
- Japan (3):
  - Reserch site, Kanto
  - Reserch site, Kinki
  - Reserch site, Tōhoku

REFERENCES:
- [Result] Kadowaki T, Inagaki N, Kondo K, Nishimura K, Kaneko G, Maruyama N, Nakanishi N, Gouda M, Iijima H, Watanabe Y. Efficacy and safety of teneligliptin added to canagliflozin monotherapy in Japanese patients with type 2 diabetes mellitus: A multicentre, randomized, double-blind, placebo-controlled, parallel-group comparative study. Diabetes Obes Metab. 2018 Feb;20(2):453-457. doi: 10.1111/dom.13079. Epub 2017 Sep 15. PMID 28786530

RESULTS

PARTICIPANT FLOW:
Groups:
- Teneligliptin+Canagliflozin: Teneligliptin for 24 weeks in combination with Canagliflozin
- Placebo+Canagliflozin: Placebo for 24 weeks in combination with Canagliflozin
Period: Overall Study
Arm/Group | Teneligliptin+Canagliflozin | Placebo+Canagliflozin
Started | 77 | 77
Completed | 73 | 66
Not Completed | 4 | 11
Not completed — Adverse Event | 0 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Conflict with the stopping criteria | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teneligliptin+Canagliflozin | Placebo+Canagliflozin | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 66 | 61 | 127
  >=65 years | 11 | 16 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 32
  Male | 64 | 58 | 122

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percentage of Glycated Hemoglobin (HbA1c)
Description: The change from baseline in percentage of HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 24.
Time Frame: Baseline, 24 Weeks
Population: Full analysis set, last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Teneligliptin+Canagliflozin | Placebo+Canagliflozin
Number analyzed (Participants) | 77 | 77
percentage of HbA1c | -0.94 (0.08) | 0.00 (0.08)
Statistical Analysis 1: Comparison: Teneligliptin+Canagliflozin vs Placebo+Canagliflozin; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -0.94, 95% CI 2-sided [-1.16 to -0.72], Standard Error of Mean 0.11

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Level
Description: The change from baseline in fasting plasma glucose level collected at Week 24.
Time Frame: Baseline, 24 Weeks
Population: Full analysis set, last observation carried forward. Outcome measure for one patient was not assessed at a certain timepoint due to dropout.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Teneligliptin+Canagliflozin | Placebo+Canagliflozin
Number analyzed (Participants) | 77 | 76
mg/dL | -5.6 (2.7) | 10.0 (2.8)
Statistical Analysis 1: Comparison: Teneligliptin+Canagliflozin vs Placebo+Canagliflozin; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -15.6, 95% CI 2-sided [-23.3 to -7.9], Standard Error of Mean 3.9

3. Secondary Outcome: Percentage Change in Body Weight From Baseline
Description: The percentage change from baseline in body weight collected at Week 24.
Time Frame: Baseline, 24 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teneligliptin+Canagliflozin | Placebo+Canagliflozin
Number analyzed (Participants) | 77 | 76
percent change | 0.09 (0.29) | -1.34 (0.29)
Statistical Analysis 1: Comparison: Teneligliptin+Canagliflozin vs Placebo+Canagliflozin; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = 1.43, 95% CI 2-sided [0.63 to 2.23], Standard Error of Mean 0.41

4. Secondary Outcome: Change From Baseline in the AUC(0-2h) for Postprandial Plasma Glucose (PPG)
Description: The change from Baseline in AUC(0-2h) for Postprandial Plasma Glucose collected at Week 24.
Time Frame: 0, 0.5, 1 and 2 hour postprandial, at Baseline and 24 Weeks
Population: Full analysis set. Outcome measure for one patient was not assessed at a certain timepoint due to dropout.
Measure: Least Squares Mean (Standard Error); unit: hour*mg/dL
Arm/Group | Teneligliptin+Canagliflozin | Placebo+Canagliflozin
Number analyzed (Participants) | 73 | 65
hour*mg/dL | -50.2 (6.3) | 5.7 (6.7)
Statistical Analysis 1: Comparison: Teneligliptin+Canagliflozin vs Placebo+Canagliflozin; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -55.9, 95% CI 2-sided [-74.1 to -37.6], Standard Error of Mean 9.2

5. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose Level
Description: The change from baseline in 2-hour postprandial plasma glucose level collected at Week 24.
Time Frame: 2 Hours Postprandial, at Baseline and 24 Weeks
Population: Full analysis set. Outcome measure for one patient was not assessed at a certain timepoint due to dropout.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Teneligliptin+Canagliflozin | Placebo+Canagliflozin
Number analyzed (Participants) | 73 | 65
mg/dL | -35.3 (4.3) | 2.3 (4.5)
Statistical Analysis 1: Comparison: Teneligliptin+Canagliflozin vs Placebo+Canagliflozin; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -37.6, 95% CI 2-sided [-49.9 to -25.2], Standard Error of Mean 6.2

ADVERSE EVENTS:
Arm/Group | Teneligliptin+Canagliflozin | Placebo+Canagliflozin
Serious Adverse Events (participants affected / at risk) | 1/77 | 2/77
Other Adverse Events (participants affected / at risk) | 15/77 | 8/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin+Canagliflozin (N=77) | Placebo+Canagliflozin (N=77)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin+Canagliflozin (N=77) | Placebo+Canagliflozin (N=77)
Nasopharyngitis (Infections and infestations) | 12 | 8
Upper respiratory tract infection (Infections and infestations) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other